CLINICAL TRIAL: NCT06643806
Title: Implementation of a Peer Leader-facilitated Dyadic Intervention to Decrease Cardiovascular Disease Risk Among First Generation Asian Indian Immigrants
Brief Title: Implementation of a Peer Leader-facilitated Dyadic Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Karen T. D'Alonzo PhD RN APN-cc., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2024002046; 1P50MD017356-01 (NIH)
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes Mellitus in Obese; Hyperlipidemias
Keywords: Community based participatory research; Asian Indian immigrants; Acculturation stress
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial of 12 week intervention.
Who Masked: Participant
Masking Description: We will attempt to enforce community level blinding/masking in this study, but other forms of blinding/masking are not entirely possible in a cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Twenty marital dyads from the site randomly assigned as the intervention site(s) will receive the 12- week peer leader-facilitated dyadic intervention. Topics over the 12 week intervention will address stress management, family history and genetic risk, dietary habits, physical activity and social support/community engagement.
  Interventions: Behavioral: CHAI dyad study
- Control (Active Comparator): Twenty dyads from the site randomly assigned as the "usual care" control group site will receive a basic cardiovascular lifestyle modification program. This program will be similar to a classic cardiac rehabilitation program and will consist of diet, physical activity and medical management.
  Interventions: Behavioral: CHAI dyad study

INTERVENTIONS:
Behavioral: CHAI dyad study — In the CHAI (Cardiovascular Health among Asian Indian immigrants) Dyad study, we plan to Implement and pilot test a peer leader-facilitated 12-week dyadic intervention to decrease CVD risk among first generation AI immigrants;

SUMMARY:
This Pilot Study Large Application builds upon the results of our prior work to 1) Implement and pilot test a peer leader-facilitated 12-week dyadic intervention (Community Health among Asian Indian immigrants (CHAI) Dyad study) using a cluster randomization design, to decrease CVD risk among first generation AI immigrants; and 2) Assess the feasibility/acceptability of a full-scale intervention. Twenty marital dyads from the site randomly assigned as the intervention site will receive the 12- week peer leader-facilitated dyadic intervention, while 20 dyads from the site randomly assigned as the "usual care" control group site will receive a basic cardiovascular lifestyle modification program. Both groups will meet weekly (90 min. classes) for 12 weeks in a hybrid format (a combination of face to face and remote learning). The intervention is designed to address factors that we identified in our previous study as contributing to a syndemic of cardiovascular disease among AI immigrants including acculturation stress, family history and genetic risk, physical inactivity, as well as a high fat, high-carbohydrate, high-calorie diet.

DETAILED DESCRIPTION:
Asian Indian (AI) immigrants, the second largest immigrant group in the US, have a high prevalence of abdominal obesity and premature cardiovascular disease (CVD). Despite ample epidemiological evidence of the need to reduce CVD risk in AIs, few published interventions have addressed this population, primarily focusing on dietary measures and promotion of physical activity, and none of these address immigrant AIs.

This Pilot Study Large Application builds upon the results of our prior work to 1) Implement and pilot test a peer leader-facilitated 12-week dyadic intervention (Community Health among Asian Indian immigrants (CHAI) Dyad study) using a cluster randomization design, to decrease CVD risk among first generation AI immigrants; and 2) Assess the feasibility/acceptability of a full-scale intervention. Twenty marital dyads from the site randomly assigned as the intervention site will receive the 12- week peer leader-facilitated dyadic intervention, while 20 dyads from the site randomly assigned as the "usual care" control group site will receive a basic cardiovascular lifestyle modification program. Both groups will meet weekly (90 min. classes) for 12 weeks in a hybrid format (a combination of face to face and remote learning). The intervention is designed to address factors that we identified in our previous study as contributing to a syndemic of cardiovascular disease among AI immigrants including acculturation stress, family history and genetic risk, physical inactivity, as well as a high fat, high-carbohydrate, high-calorie diet.

Unlike a hypothesis generating study, a pilot study is designed to assess the feasibility/accessibility of an approach to be used in a larger scale study. The following research questions are designed to address feasibility and accessibility of this pilot cluster randomized controlled trial intervention:

Q1 Can the target population of AI immigrant dyads be recruited from faith-based or AI community-based organizations in Central and Northern NJ? Q2 Can the target population of AI immigrant dyads be randomized in a cluster randomized controlled trial? Q3 Can the target population of AI immigrant dyads be retained? Q4 Can the treatments be delivered per protocol? Q5 Will AI immigrant dyads adhere to the treatment protocol? Q6 Are the treatment conditions of the intervention acceptable to AI immigrant dyads?

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling first generation Asian Indian (AI) immigrants (in marital dyads) between the ages of 18-70 years of age who can read and write English and are technology literate.

Exclusion Criteria:

* AIs not in a marital dyad, those below the age of 20 or above 70 years or those born in the US or visiting the US from India.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-report of gender identity.
Enrollment: 80 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Risk of CVD | 13 weeks
  Measured by the QRISK3

SECONDARY OUTCOMES:
Acculturation stress | 13 weeks
  Measured by the Riverside Acculturation Stress Inventory
Perceived stress | 13 weeks
  Measured by the Perceived Stress Scale
Body composition | 13 weeks
  BMI (weight and height will be combined to report BMI in kg/m^2)
waist circumference | 13 weeks
  Body composition
Hemoglobin A1c | 13 weeks
  Measure of glucose control
Lipid panel | 13 weeks
  Total cholesterol, HDL, LDL, triglycerides
Inflammation | 13 weeks
  C-reactive protein
Genetic risk of CVD | 13 weeks
  Lipoprotein a

OTHER OUTCOMES:
Community support | 13 weeks
  Perceived community support questionnaire
Salivary cortisol | 13 weeks
  three specimens (upon rising, one-half hour later and at bedtime)
Physical activity | 13 weeks
  NASA JSC physical activity scale
dietary intake | 13 weeks
  3 day dietary diary

CONTACTS AND LOCATIONS:
Overall Officials: Karen T D'Alonzo, PhD, Principal Investigator — Rutgers, The State University of New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available immediately after publication with no end date.
Access Criteria: Data will be made available indefinitely at a specific link (to be determined)